CLINICAL TRIAL: NCT04559659
Title: Study of the Relationship Between Respiratory Muscle Strenght, Peripheral Muscle Blood Flow and Gait Speed in the Elderly
Brief Title: Relationship Between Respiratory Muscle Strenght, Peripheral Muscle Blood Flow and Gait Speed in the Elderly
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Principal Investigator, Luciana Diniz Nagem Janot Matos, PhD, Hospital Israelita Albert Einstein
Other Study IDs: 3157-17
Record Dates: First submitted 2018-07-27; First posted 2020-09-23 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Age Problem
Keywords: blood flow velocity; aging; respiratory pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Respiratory muscle strength — Pimax and Pmax will be performed according to the (ATS) and (ERS). A Manovacuometer (Analog M 120, GlobalMed) with a range between 0-120cmH2O will be used. The elderly should undergo forced inspiration after maximal expiration and forced expiration after maximal inspiration through a mouthpiece with a hole to prevent closure of the glottis to evaluate Pimax and Pmax. The elderly should sustain the inspiration for 1 second. Three measurements will be performed, with a one-minute interval between them, with less difference equal to 10% between them, the higher value will be used.

SUMMARY:
The pourpose of this study is to verify if have relationship between respiratory muscle strenght, peripheral muscle blood flow and gait speed in the elderly.

DETAILED DESCRIPTION:
The hypothesis of this study is that elderly with inspiratory muscle weakness will present lower peripheral blood flow and consequently lower walking speed. The main aim of the study is to verify if the peripheral muscular blood flow in the elderly is different between patients with and without decrease in inspiratory muscle strength. As secondary objectives, it will be evaluated the correlation between inspiratory muscle strength and gait speed and quality of life, as well as gait speed and peripheral muscle blood flow. Fifty elderly patients of both sexes, over 65 years, from Vila Mariana Einstein Outpatient Clinic and Cora Residencial Senior, will be included to evaluate Maximum Inspiratory Pressure (Pimáx), Maximum Expiratory Pressure (Pemáx), Spirometry (FVC, PF, FEV1), 4.6m Walk Test, Quality of life for the elderly (WHOQOL old), Mini Mental Test, Body Mass Index (BMI) and peripheral muscle blood flow by venous occlusion plethysmography.

ELIGIBILITY:
Inclusion Criteria: Elderly of both sexes, over 65 years old

-

Exclusion Criteria:

* Mini Mental Test <24
* Morse ≥ 51
* Clinical instability, according to medical assessment • Structural heart disease, with ejection fraction <50% and chronic lung diseases with FEV1 <50% predicted,
* Neurological, orthopedic, or neuromuscular diseases that prevent the performance of evaluations
* Smokers or ex-smokers <5 years

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly of both sexes, over 65 years old, with and without inspiratory muscle weakness.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Peripheral muscle blood flow, gait speed and handgrip strength | Day 1
  Check if there is a correlation between peripheral muscle blood flow, gait speed and handgrip strength and if this association is mediated by inspiratory muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana D Janot, doctor, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- RIAE Vila Mariana, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cebria I Iranzo MD, Arnall DA, Igual Camacho C, Tomas JM, Melendez JC. Physiotherapy intervention for preventing the respiratory muscle deterioration in institutionalized older women with functional impairment. Arch Bronconeumol. 2013 Jan;49(1):1-9. doi: 10.1016/j.arbres.2012.07.007. Epub 2012 Sep 19. English, Spanish. PMID 22999331
- [Background] Ribeiro JP, Chiappa GR, Callegaro CC. The contribution of inspiratory muscles function to exercise limitation in heart failure: pathophysiological mechanisms. Rev Bras Fisioter. 2012 Jul-Aug;16(4):261-7. doi: 10.1590/s1413-35552012005000034. Epub 2012 Jul 17. English, Portuguese. PMID 22801449
- [Background] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Background] Cosa D, Goncalves HA, Lima LP, Ike D, Cancelliero KM, Montebelo MI. New reference values for maximal respiratory pressures in the Brazilian population: corrections. J Bras Pneumol. 2010 Sep-Oct;36(5):667. doi: 10.1590/s1806-37132010000500021. No abstract available. English, Portuguese. PMID 21085835
- [Background] Ritti-Dias RM, Cucato GG, de Mello Franco FG, Cendoroglo MS, Nasri F, Monteiro-Costa ML, de Carvalho JA, de Matos LD. Peak expiratory flow mediates the relationship between handgrip strength and timed up and go performance in elderly women, but not men. Clinics (Sao Paulo). 2016 Sep;71(9):517-20. doi: 10.6061/clinics/2016(09)06. PMID 27652833
- [Background] Dumurgier J, Elbaz A, Ducimetiere P, Tavernier B, Alperovitch A, Tzourio C. Slow walking speed and cardiovascular death in well functioning older adults: prospective cohort study. BMJ. 2009 Nov 10;339:b4460. doi: 10.1136/bmj.b4460. PMID 19903980
- [Background] Enright PL, Kronmal RA, Manolio TA, Schenker MB, Hyatt RE. Respiratory muscle strength in the elderly. Correlates and reference values. Cardiovascular Health Study Research Group. Am J Respir Crit Care Med. 1994 Feb;149(2 Pt 1):430-8. doi: 10.1164/ajrccm.149.2.8306041.
- [Background] Vaz Fragoso CA, Beavers DP, Hankinson JL, Flynn G, Berra K, Kritchevsky SB, Liu CK, McDermott MM, Manini TM, Rejeski WJ, Gill TM; Lifestyle Interventions Independence for Elders Study Investigators. Respiratory impairment and dyspnea and their associations with physical inactivity and mobility in sedentary community-dwelling older persons. J Am Geriatr Soc. 2014 Apr;62(4):622-8. doi: 10.1111/jgs.12738. Epub 2014 Mar 17. PMID 24635756
- [Background] Fragoso CA, Gahbauer EA, Van Ness PH, Concato J, Gill TM. Peak expiratory flow as a predictor of subsequent disability and death in community-living older persons. J Am Geriatr Soc. 2008 Jun;56(6):1014-20. doi: 10.1111/j.1532-5415.2008.01687.x. Epub 2008 Apr 18. PMID 18422951
- [Background] Harms CA, Babcock MA, McClaran SR, Pegelow DF, Nickele GA, Nelson WB, Dempsey JA. Respiratory muscle work compromises leg blood flow during maximal exercise. J Appl Physiol (1985). 1997 May;82(5):1573-83. doi: 10.1152/jappl.1997.82.5.1573. PMID 9134907
- [Background] Higashi Y, Yoshizumi M. New methods to evaluate endothelial function: method for assessing endothelial function in humans using a strain-gauge plethysmography: nitric oxide-dependent and -independent vasodilation. J Pharmacol Sci. 2003 Dec;93(4):399-404. doi: 10.1254/jphs.93.399. PMID 14737008
- [Result] Buchman AS, Boyle PA, Leurgans SE, Evans DA, Bennett DA. Pulmonary function, muscle strength, and incident mobility disability in elders. Proc Am Thorac Soc. 2009 Dec 1;6(7):581-7. doi: 10.1513/pats.200905-030RM. PMID 19934353